CLINICAL TRIAL: NCT00924443
Title: A Phase II Trial of Clofarabine in Older Patients With Acute Myeloid Leukemia for Whom Intensive Chemotherapy is Not Considered Suitable
Brief Title: A Study of Clofarabine in Older Patients With Acute Myeloid Leukemia (AML) for Whom Chemotherapy Is Not Suitable
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Bioenvision (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOV-121
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myelogenous leukemia; acute myeloid leukemia; clolar; evoltra; clofarabine; untreated acute leukemia; adult acute leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clofarabine (Experimental): Clofarabine 30 mg/m^2/day intravenously over 1 hour for 5 days every 28 to 42 days (one cycle), then 20mg/m^2/day intravenously over 1 hour for 5 days every 29 to 43 days for the second and subsequent cycles, up to a maximum of 3 cycles.
  Interventions: Drug: clofarabine

INTERVENTIONS:
Drug: clofarabine
  Other Names: tradename US = Clolar; tradename EU = Evoltra

SUMMARY:
The purpose of the study is to determine if treatment of older patients indicated with untreated Acute Myeloid Leukemia (AML) who are not considered to be suitable for intensive chemotherapy, can effectively be treated with Clofarabine.

DETAILED DESCRIPTION:
Note: This clinical trial was conducted by Bioenvision Ltd. Bioenvision Ltd. was acquired by Genzyme Corporation Oct 2007.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed, written informed consent
* Have untreated AML according to World Health Organization (WHO) classification
* Male or post-menopausal female ≥ 65 years of age
* Unsuitable for intensive chemotherapy
* Be able to comply with study procedures and follow-up examination
* Male patient who are fertile agree to use and effective barrier method of birth control to avoid pregnancies
* Have adequate liver and renal function as indicated by certain laboratory values

Exclusion Criteria:

* Received previous treatment with clofarabine
* Are receiving other chemotherapy or corticosteroids (low-dose corticosteroid for pre-medication purposes are allowed)
* Have received prior treatment for leukemia. Growth factor, cytokine support, leukopheresis or hydroxyurea will be allowed but must be discontinued at least 24 hours prior to start of treatment with clofarabine
* Have a psychiatric disorder that would interfere with consent, study participation, or follow-up
* Have an active, uncontrolled systemic infection
* Are currently participating in other investigational drug studies or having received other investigational drugs within the previous 30 days
* Have symptomatic central nervous system (CNS) involvement
* Blast transformation of chronic myeloid leukemia or acute promyelocytic leukemia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-06; Primary Completion 2006-06 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (15):
- Dublin, Ireland
- Italy (2):
  - Bologna
  - Rome
- United Kingdom (12):
  - Belfast, Northern Ireland
  - Aberdeen
  - Birmingham
  - Cardiff
  - Edinburgh
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Nottingham
  - Somerset
  - Taunton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were entered into the study between 14 Jun 2004 and 14 Nov 2005. Participants were recruited from 14 of a total of 17 registered centres located in the United Kingdom (UK), Ireland and Italy. Relapse and survival data follow-up cut-off was extended to 23 May 2008.
Pre-assignment Details: A total of 69 participants were screened and enrolled. A total of 66 participants received study drug and are included in the reported results.
Groups:
- Clofarabine: Clofarabine 30 mg/m^2/day intravenously over 1 hour for 5 days every 29 to 43 days
Period: Overall Study
Arm/Group | Clofarabine
Started | 69
Full Analysis Set (Received Study Drug) | 66
Completed | 66
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics provided for Full Analysis Set (FAS) population, defined as all participants with a confirmed diagnosis of AML who received at least one dose of clofarabine
Arm/Group | Clofarabine
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 3
  Italy | 8
  United Kingdom | 55
Cytogenetics (1998) [Number; unit: participants] — Diagnostic criteria of Grimwade for younger patients
  participants
    Favourable | 0
    Intermediate | 43
    Adverse | 19
    Missing/Unknown | 4
Cytogenetics (2001) [Number; unit: participants] — Diagnostic criteria of Grimwade for older patients
  participants
    Favourable | 0
    Intermediate | 48
    Adverse | 14
    Missing/Unknown | 4
Type of Acute Myeloid Leukemia (AML) [Number; unit: participants]
  De Novo | 48
  Secondary | 16
  Missing/Unknown | 2
White Blood Cell Count (10^9/L) [Number; unit: participants]
  <25 | 57
  25-99.9 | 6
  >=100 | 3
Glomerular Filtration Rate (mL/min/1.73m^2) [Number; unit: participants]
  <=50 | 15
  >50 | 51
Number of Co-morbidities [Number; unit: participants]
  0 | 17
  1 | 23
  >1 | 26
Karnofsky Performance Status [Number; unit: participants] — Karnofsky performance scale is used by doctors to classify patient's functional impairment level. The lower the number the higher the impairment in typical daily activities by the disease.
  Typical classification examples: 100% normal with no evidence of disease, 90% able to carry on normal activity with minor signs of illness, 80% normal activity but requiring effort, 70% able to care for self but unable to work or carry on other normal activities, 60% able to care for most needs but requires occasional assistance, 50% considerable assistance and frequent medical care required, etc..
  participants
    100% | 8
    90% | 13
    80% | 24
    70% | 9
    60% | 2
    50% | 5
    20% | 2
    Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR rate was defined as the sum of the number of participants in the study population with complete remission (CR), complete remission with incomplete blood count recovery (CRi), or partial remission (PR) divided by the total number of participants in the study population.
  ORR rate was determined by assessment of morphology and blast count from bone marrow aspirates and peripheral blood performed prior to first dose and at the end of clofarabine treatment. The ORR was determined at the end of each cycle of clofarabine, and assessed using the participant's best response to clofarabine treatment.
Time Frame: At month 20
Population: The efficacy analysis was performed on the primary analysis population, the Full Analysis Set population, which consisted of all participants with a diagnosis of AML confirmed by the Investigator who received at least one dose (partial or complete) of clofarabine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 66
percentage of participants | 48 [36 to 61]

2. Secondary Outcome: Rate of Response (Complete, Complete With Incomplete Blood Count Recovery, Partial)
Description: Response was determined by assessment of morphology and blast count from bone marrow aspirates and peripheral blood performed prior to first dose and at the end of clofarabine treatment.
  Response was determined at the end of each cycle of clofarabine, and assessed using the participant's best response to clofarabine treatment.
Time Frame: At month 20
Population: The efficacy analyses were performed on the primary analysis population, the Full Analysis Set population, which consisted of all participants with a diagnosis of AML confirmed by the Investigator who received at least one dose (partial or complete) of clofarabine.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 66
percent of participants
  Complete response | 21 [12 to 33]
  Complete with incomplete blood count recovery | 23 [13 to 35]
  Partial response | 5 [1 to 13]

3. Secondary Outcome: Duration of Overall Response
Description: Duration was calculated by Kaplan-Meier estimates
Time Frame: From 20 months up to 48 months
Population: The analysis were performed on the primary analysis population, the Full Analysis Set population. Defined as the median duration of overall response (CR+CRi+PR) in participants who achieved CR, CRi or PR only
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Clofarabine
Number analyzed (Participants) | 32
days | 62 [42 to 153]

4. Secondary Outcome: Overall Survival
Description: Calculated by Kaplan-Meier estimates
Time Frame: From 20 months up to 48 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Clofarabine
Number analyzed (Participants) | 66
days | 173 [90 to 295]

5. Secondary Outcome: Duration of Complete Remission
Description: Duration was calculated by Kaplan- Meier estimates
Time Frame: From 20 months up to 48 months
Population: The analysis were performed on the primary analysis population, the Full Analysis Set population. Defined as the median duration of participants who achieved CR+CRi only
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
days | 63 [43 to 168]

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after study completion (20 months)
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator (""number of affected participants"") of both adverse event tables.
Groups:
- Clofarabine: Clofarabine 30 mg/m^2/day intravenously over 1 hour for 5 days every 28 to 42 days(one cycle) and 20 mg/m^2/day intravenously over 1 hour for 5 days every 29 to 43 days for second and subsequent cycles,up to a maximum of 3 cycles.
Arm/Group | Clofarabine
Serious Adverse Events (participants affected / at risk) | 40/66
Other Adverse Events (participants affected / at risk) | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine (N=66)
ANAEMIA (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 1
PLATELET DISORDER (Blood and lymphatic system disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 4
PERICARDIAL EFFUSION (Cardiac disorders) | 1
HYPOPITUITARISM (Endocrine disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 2
DISEASE PROGRESSION (General disorders) | 1
OEDEMA (General disorders) | 1
PYREXIA (General disorders) | 2
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1
BACTERAEMIA (Infections and infestations) | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1
CATHETER RELATED INFECTION (Infections and infestations) | 1
CENTRAL LINE INFECTION (Infections and infestations) | 1
ENCEPHALITIS HERPES (Infections and infestations) | 1
INFECTION (Infections and infestations) | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
NEUTROPENIC SEPSIS (Infections and infestations) | 17
PNEUMONIA (Infections and infestations) | 4
RESPIRATORY TRACT INFECTION FUNGAL (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 5
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
URINE OUTPUT DECREASED (Investigations) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
PITUITARY TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 3
HEADACHE (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
UNRESPONSIVE TO PAIN STIMULI (Nervous system disorders) | 1
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 7
RENAL IMPAIRMENT (Renal and urinary disorders) | 2
RENAL INSUFFICIENCY (Renal and urinary disorders) | 5
RASH (Skin and subcutaneous tissue disorders) | 2
SKIN DESQUAMATION (Skin and subcutaneous tissue disorders) | 1
HYPOTENSION (Vascular disorders) | 1
THROMBOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine (N=66)
ANAEMIA (Blood and lymphatic system disorders) | 22
COAGULOPATHY (Blood and lymphatic system disorders) | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 19
PANCYTOPENIA (Blood and lymphatic system disorders) | 1
SPLENOMEGALY (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 32
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 4
PALPITATIONS (Cardiac disorders) | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1
HYPOTHALAMO-PITUITARY DISORDERS (Endocrine disorders) | 1
HYPOTHYROIDISM (Endocrine disorders) | 1
EYE PAIN (Eye disorders) | 1
EYE REDNESS (Eye disorders) | 1
HETEROPHORIA (Eye disorders) | 1
KERATOCONJUNCTIVITIS SICCA (Eye disorders) | 2
LACRIMATION INCREASED (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 13
CHEILITIS (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 27
DIARRHOEA (Gastrointestinal disorders) | 40
DRY MOUTH (Gastrointestinal disorders) | 6
DYSPEPSIA (Gastrointestinal disorders) | 5
DYSPHAGIA (Gastrointestinal disorders) | 1
ERUCTATION (Gastrointestinal disorders) | 1
FAECALOMA (Gastrointestinal disorders) | 1
FLATULENCE (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 1
GLOSSODYNIA (Gastrointestinal disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 1
LOOSE STOOLS (Gastrointestinal disorders) | 2
MELAENA (Gastrointestinal disorders) | 2
MOUTH ULCERATION (Gastrointestinal disorders) | 6
NAUSEA (Gastrointestinal disorders) | 44
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1
ORAL MUCOSAL BLISTERING (Gastrointestinal disorders) | 1
ORAL MUCOSAL PETECHIAE (Gastrointestinal disorders) | 1
ORAL PAIN (Gastrointestinal disorders) | 5
RECTAL PROLAPSE (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 5
SWOLLEN TONGUE (Gastrointestinal disorders) | 1
TONGUE BLISTERING (Gastrointestinal disorders) | 1
TONGUE COATED (Gastrointestinal disorders) | 3
TONGUE ULCERATION (Gastrointestinal disorders) | 1
TOOTHACHE (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 37
ASTHENIA (General disorders) | 7
CATHETER RELATED COMPLICATION (General disorders) | 14
CATHETER SITE INFLAMMATION (General disorders) | 1
CHEST DISCOMFORT (General disorders) | 1
CHEST PAIN (General disorders) | 11
FATIGUE (General disorders) | 16
GAIT ABNORMAL (General disorders) | 2
GENERALISED OEDEMA (General disorders) | 1
INFLUENZA LIKE ILLNESS (General disorders) | 2
LOCALISED OEDEMA (General disorders) | 1
MASS (General disorders) | 1
MUCOSAL INFLAMMATION (General disorders) | 2
OEDEMA (General disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 12
PAIN (General disorders) | 3
PITTING OEDEMA (General disorders) | 1
PYREXIA (General disorders) | 24
RIGORS (General disorders) | 7
TENDERNESS (General disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1
HEPATOTOXICITY (Hepatobiliary disorders) | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 4
HYPERSENSITIVITY (Immune system disorders) | 2
ANAL INFECTION (Infections and infestations) | 1
BACTERIAL INFECTION (Infections and infestations) | 2
BACTERIAL SEPSIS (Infections and infestations) | 2
CELLULITIS (Infections and infestations) | 7
CENTRAL LINE INFECTION (Infections and infestations) | 11
CLOSTRIDIAL INFECTION (Infections and infestations) | 1
CLOSTRIDIUM COLITIS (Infections and infestations) | 1
FUNGAL INFECTION (Infections and infestations) | 1
GASTROINTESTINAL CANDIDIASIS (Infections and infestations) | 1
GENITAL INFECTION FEMALE (Infections and infestations) | 1
HERPES SIMPLEX (Infections and infestations) | 3
HERPES VIRUS INFECTION (Infections and infestations) | 1
INFECTION (Infections and infestations) | 9
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4
NASOPHARYNGITIS (Infections and infestations) | 1
NEUTROPENIC INFECTION (Infections and infestations) | 2
NEUTROPENIC SEPSIS (Infections and infestations) | 3
ORAL CANDIDIASIS (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 3
PNEUMONIA FUNGAL (Infections and infestations) | 2
RHINITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 5
URINARY TRACT INFECTION (Infections and infestations) | 2
VANCOMYCIN-RESISTANT ENTEROCOCCAL INFECTION (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 2
BLISTER (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 4
FALL (Injury, poisoning and procedural complications) | 3
MEDICAL DEVICE DISCOMFORT (Injury, poisoning and procedural complications) | 1
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 3
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 21
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 15
BACTERIA BLOOD IDENTIFIED (Investigations) | 1
BACTERIA STOOL IDENTIFIED (Investigations) | 1
BLOOD ALBUMIN DECREASED (Investigations) | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 5
BLOOD BICARBONATE DECREASED (Investigations) | 4
BLOOD BILIRUBIN INCREASED (Investigations) | 6
BLOOD CALCIUM DECREASED (Investigations) | 3
BLOOD CREATININE (Investigations) | 1
BLOOD CREATININE ABNORMAL (Investigations) | 2
BLOOD CREATININE DECREASED (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 8
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 9
BLOOD MAGNESIUM (Investigations) | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 2
BLOOD MAGNESIUM INCREASED (Investigations) | 2
BLOOD PHOSPHORUS DECREASED (Investigations) | 3
BLOOD PHOSPHORUS INCREASED (Investigations) | 1
BLOOD POTASSIUM DECREASED (Investigations) | 11
BLOOD PRESSURE DECREASED (Investigations) | 1
BLOOD SODIUM DECREASED (Investigations) | 3
BLOOD SODIUM INCREASED (Investigations) | 1
BLOOD UREA DECREASED (Investigations) | 1
BLOOD UREA INCREASED (Investigations) | 10
BODY TEMPERATURE INCREASED (Investigations) | 1
CARDIAC MURMUR (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 6
HEART RATE IRREGULAR (Investigations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 3
NEUTROPHIL COUNT DECREASED (Investigations) | 1
PLATELET COUNT DECREASED (Investigations) | 6
PROTEIN TOTAL DECREASED (Investigations) | 2
PROTHROMBIN TIME PROLONGED (Investigations) | 1
TROPONIN T INCREASED (Investigations) | 1
URINE OUTPUT DECREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 3
WEIGHT INCREASED (Investigations) | 4
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2
ACIDOSIS (Metabolism and nutrition disorders) | 2
ANOREXIA (Metabolism and nutrition disorders) | 10
DECREASED APPETITE (Metabolism and nutrition disorders) | 17
DEHYDRATION (Metabolism and nutrition disorders) | 5
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 2
FLUID OVERLOAD (Metabolism and nutrition disorders) | 2
GOUT (Metabolism and nutrition disorders) | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 6
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 11
HYPOKALAEMIA (Metabolism and nutrition disorders) | 23
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 5
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7
BURNING SENSATION (Nervous system disorders) | 2
CENTRAL NERVOUS SYSTEM INFLAMMATION (Nervous system disorders) | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 11
DYSARTHRIA (Nervous system disorders) | 1
DYSGEUSIA (Nervous system disorders) | 3
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 14
HYPERAESTHESIA (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 1
LETHARGY (Nervous system disorders) | 7
PARAESTHESIA (Nervous system disorders) | 1
POLYNEUROPATHY (Nervous system disorders) | 1
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1
SOMNOLENCE (Nervous system disorders) | 1
SPEECH DISORDER (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 3
SYNCOPE VASOVAGAL (Nervous system disorders) | 3
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
AGITATION (Psychiatric disorders) | 5
ANXIETY (Psychiatric disorders) | 7
CONFUSIONAL STATE (Psychiatric disorders) | 9
DEPRESSED MOOD (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 2
DISORIENTATION (Psychiatric disorders) | 1
EMOTIONAL DISTRESS (Psychiatric disorders) | 1
HALLUCINATION (Psychiatric disorders) | 6
INSOMNIA (Psychiatric disorders) | 9
PANIC ATTACK (Psychiatric disorders) | 1
PSYCHIATRIC SYMPTOM (Psychiatric disorders) | 1
SLEEP DISORDER (Psychiatric disorders) | 1
DYSURIA (Renal and urinary disorders) | 2
HAEMATURIA (Renal and urinary disorders) | 5
OLIGURIA (Renal and urinary disorders) | 1
POLLAKIURIA (Renal and urinary disorders) | 1
RENAL COLIC (Renal and urinary disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3
RENAL IMPAIRMENT (Renal and urinary disorders) | 7
RENAL INSUFFICIENCY (Renal and urinary disorders) | 2
RENAL TUBULAR DISORDER (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 4
BALANITIS (Reproductive system and breast disorders) | 1
PENIS DISORDER (Reproductive system and breast disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1
APNOEIC ATTACK (Respiratory, thoracic and mediastinal disorders) | 1
CAPILLARY LEAK SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 13
CRACKLES LUNG (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 1
LUNG CREPITATION (Respiratory, thoracic and mediastinal disorders) | 6
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 8
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 6
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 3
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 3
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 7
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 3
LOCALISED SKIN REACTION (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
PALMAR ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 7
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1
PURPURA (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 29
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 3
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 3
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1
INADEQUATE DIET (Social circumstances) | 1
FLUSHING (Vascular disorders) | 2
HAEMORRHAGE (Vascular disorders) | 2
HYPERTENSION (Vascular disorders) | 7
HYPOTENSION (Vascular disorders) | 11
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
PETECHIAE (Vascular disorders) | 5
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI) and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed. In multi-site studies, PI can publish after sponsor publishes or 18 months after study completion. PI gives sponsor a draft 60 days before publication. Sponsor can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application.